CLINICAL TRIAL: NCT03712904
Title: Phase II Randomized Trial of Stereotactic Radiotherapy (SRT) Followed by Intravitreal Aflibercept Injection for Patients With Ocular Melanoma
Brief Title: Stereotactic Body Radiation Therapy and Aflibercept in Treating Patients With Uveal Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18P.457; JT 11801 (Other: JeffTrial Number)
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Radiosurgery; aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- A. Stereotactic body radiation therapy, ziv-aflibercept (Experimental): Patients undergo stereotactic body radiation therapy over 5 fractions every other week day during days 1-10. Patients then receive ziv-aflibercept IVI on the last day of radiation therapy and then every 2 months for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Stereotactic Body Radiation Therapy
- B. Stereotactic body radiation therapy, ziv-aflibercept (Experimental): Patients undergo stereotactic body radiation therapy as in arm A. Patients then receive ziv-aflibercept IVI on the last day of radiation therapy and then every 4 months for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Ziv-Aflibercept

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Undergo radiation
  Other Names: SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: A. Stereotactic body radiation therapy, ziv-aflibercept
Biological: Ziv-Aflibercept — Given IV
  Other Names: 724770; 862111-32-8; AVE0005; Eylea; Vascular Endothelial Growth Factor Trap
  Arms: B. Stereotactic body radiation therapy, ziv-aflibercept

SUMMARY:
This phase II trial studies how well stereotactic body radiation therapy and aflibercept work in treating patients with uveal melanoma. Stereotactic body radiation therapy is a specialized radiation therapy that sends x-rays directly to the tumor using smaller doses over several days and may cause less damage to normal tissue. Aflibercept may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving stereotactic body radiation therapy followed by aflibercept may work better in treating patients with uveal melanoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the percentage of patients able to successfully complete their prescribed treatment of radiation and intravitreal ziv-aflibercept (aflibercept) injection (IAI) with an acceptable level of toxicity.

SECONDARY OBJECTIVES:

I. To assess for reduction in the incidence of 2-year rates of radiation maculopathy, radiation papillopathy, functional vision preservation, radiation glaucoma, and to assess 2-year local control and progression-free survival.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form or have a Legally Authorized Representative (LAR) who can give consent
* Willing to comply with all study procedures and be available for the duration of the study
* Must be a candidate for radiation therapy
* Karnofsky performance status (KPS) >= 60
* Diagnosed with uveal melanoma either clinically or pathologically on biopsy
* Uveal melanoma of one eye only
* Localized uveal melanoma, with no evidence of metastasis
* Women of childbearing potential must have a negative urine or serum pregnancy test within 14 days prior to enrollment

Exclusion Criteria:

* Tumor thickness more than 14 mm as measured by ultrasound
* Active collagen vascular disease
* Any contraindication to intravitreal injections including: elevated intraocular pressure, ocular or periocular infection, active intraocular inflammation, or other determined by treating physician
* Known allergic reactions to components of intravitreal Aflibercept
* Patients with known hypercoagulable syndromes
* Prior radiation to the eye or brain
* Life expectancy less than 6 months
* Blind in both eyes
* Patients unable to receive contrast enhanced brain magnetic resonance imaging (MRI)
* Deaf in both ears
* Patients have hypersensitivity to intravitreal Aflibercept
* Patients is on or within 1 month of systemic anti-VEGF treatment
* Patients who are candidates for brachytherapy
* Patients for whom enucleation is standard of care
* Pregnancy or active breastfeeding. Sexually active men or women of childbearing potential who are unwilling to practice adequate contraception prior to the initial dose/start of the first treatment, during the study, and for at least 3 months after the last dose. Adequate contraceptive measures include stable use of oral contraceptives or other prescription pharmaceutical contraceptives for 2 or more menstrual cycles prior to screening; intrauterine device; bilateral tubal ligation; vasectomy; condom plus contraceptive sponge, foam, or jelly, or diaphragm plus contraceptive sponge, foam, or jelly

  * Contraception is not required for men with documented vasectomy
  * Postmenopausal women must be amenorrheic for at least 12 months in order not to be considered of childbearing potential. Pregnancy testing and contraception are not required for women with documented hysterectomy or tubal ligation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wenyin Shi, MD, PhD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | A. Stereotactic Body Radiation Therapy, Ziv-aflibercept | B. Stereotactic Body Radiation Therapy, Ziv-aflibercept
Started | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — progression/eye removed before 2 years (unable to complete testing) | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A. Stereotactic Body Radiation Therapy, Ziv-aflibercept | B. Stereotactic Body Radiation Therapy, Ziv-aflibercept | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 2 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Percent of patients who experience Common Terminology Criteria for Adverse Events (CTCAE) v5.0 grade ≥3 toxicity related to SRT and/or intravitreal Aflibercept.
Time Frame: Up to approximately 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | A. Stereotactic Body Radiation Therapy, Ziv-aflibercept | B. Stereotactic Body Radiation Therapy, Ziv-aflibercept
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

2. Secondary Outcome: Radiation Maculopathy Rate Defined as Ophthalmoscopic Detection of Macular Edema Perivascular Sheathing
Description: Will be estimated separately in each arm with the corresponding exact binomial 90% confidence interval.
Time Frame: At 2 years
Population: No participants were evaluable for this outcome. One participant withdrew consent, one experienced disease progression requiring eye removal prior to the assessment time point, and one died before reaching the two year mark. Subject who died was no longer a patient at the institution and their death was found through obituary search.
Arm/Group | A. Stereotactic Body Radiation Therapy, Ziv-aflibercept | B. Stereotactic Body Radiation Therapy, Ziv-aflibercept
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Radiation Papillopathy Rate Defined as Ophthalmoscopic Detection of Peripapillary Encircling Nerve Fiber Layer Infarction
Description: Will be estimated separately in each arm with the corresponding exact binomial 90% confidence interval.
Time Frame: At 2 years
Population: as for outcome 2
Arm/Group | A. Stereotactic Body Radiation Therapy, Ziv-aflibercept | B. Stereotactic Body Radiation Therapy, Ziv-aflibercept
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The PI will follow adverse events with start dates occurring any time after informed consent is obtained until 7 (for non-serious AEs) or 30 days (for SAEs) after the last day of study participation. Up to approximately 6 months.
Description: Adverse events will be graded for severity according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
Arm/Group | A. Stereotactic Body Radiation Therapy, Ziv-aflibercept | B. Stereotactic Body Radiation Therapy, Ziv-aflibercept
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 1/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A. Stereotactic Body Radiation Therapy, Ziv-aflibercept (N=1) | B. Stereotactic Body Radiation Therapy, Ziv-aflibercept (N=2)
Retinal detachment - Grade 3 (Eye disorders) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) — participant death was identified via obituary search. No cause of death found.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A. Stereotactic Body Radiation Therapy, Ziv-aflibercept (N=1) | B. Stereotactic Body Radiation Therapy, Ziv-aflibercept (N=2)
Allergic Rhinitis - Grade 1 (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Atrial Fibrillation - Grade 3 (Cardiac disorders) | 1 (1) | 0 (0)
Bloating - Grade 1 (General disorders) | 0 (0) | 1 (1)
Blurred Vision - Grade 1 (Eye disorders) | 0 (0) | 2 (2)
Cardiac Myopathy - Grade 1 (Cardiac disorders) | 1 (1) | 0 (0)
Cataract - Grade 1 (Eye disorders) | 1 (1) | 0 (0)
Chronic Kidney Disease - Grade 1 (Hepatobiliary disorders) | 0 (0) | 1 (1)
Coronary Artery Disease - Grade 1 (Cardiac disorders) | 0 (0) | 1 (1)
Dyspnea - Grade 1 (Vascular disorders) | 0 (0) | 1 (1)
Episcleritis - eye - Grade 1 (Eye disorders) | 1 (1) | 0 (0)
Erythma - face - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eye Hemorrhage - Grade 2 (Eye disorders) | 0 (0) | 2 (2)
Eye Pain - Grade 1 (Eye disorders) | 0 (0) | 2 (2)
Fatigue - Grade 1 (General disorders) | 0 (0) | 1 (1)
Flashing lights - eye - Grade 1 (Eye disorders) | 1 (1) | 0 (0)
Floaters - Eye - Grade 1 (Eye disorders) | 1 (1) | 0 (0)
Focal dissection in right hepatic artery - Grade 1 (Vascular disorders) | 0 (0) | 1 (1)
Foreign body sensation - eye - Grade 1 (Eye disorders) | 1 (1) | 0 (0)
Hearing impairment - Grade 1 (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hernia - Grade 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hyperglycemia - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypertension - Grade 3 (Vascular disorders) | 1 (1) | 2 (2)
Impaired fasting glucose - Grade 1 (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Impaired Hearing - Grade 1 (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hyperkalemia - Grade 1 (Hepatobiliary disorders) | 0 (0) | 1 (1)
Left Eye Buckle - Grade 1 (Eye disorders) | 0 (0) | 1 (1)
Left eye superior arc worse - Grade 1 (Eye disorders) | 0 (0) | 1 (1)
Microcytic anemia - Grade 1 (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Myelodysplastic Syndrome - Grade 1 (Cardiac disorders) | 0 (0) | 1 (1)
Nuclear sclerosis - both eyes - Grade 1 (Eye disorders) | 1 (1) | 0 (0)
Osteoarthritis - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain - Back - Grade 1 (General disorders) | 1 (1) | 1 (1)
Periorbital changes - Grade 1 (Eye disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Photophobia - Grade 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Redness - Eye - Grade 1 (Eye disorders) | 1 (1) | 0 (0)
Renal insufficiency - Grade 1 (Hepatobiliary disorders) | 0 (0) | 1 (1)
Retinal detachment - Grade 2 (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment - Grade 3 (Eye disorders) | 1 (1) | 0 (0)
Right Eye Cystoid Macular Edema - Grade 1 (Eye disorders) | 0 (0) | 1 (1)
Spinal stenosis - lumbar region - Grade 1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Subretinal Fluid - Grade 1 (Eye disorders) | 0 (0) | 2 (2)
Swelling - Eye - Grade 1 (General disorders) | 1 (1) | 0 (0)
Tinnitus - Grade 1 (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vision decreased - Grade 1 (Eye disorders) | 1 (1) | 0 (0)
Visual field defect - Grade 1 (Eye disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/04/NCT03712904/Prot_SAP_000.pdf